CLINICAL TRIAL: NCT04442165
Title: Characterising Transmission of SARS-CoV-2 in a Peri-urban Population in Mozambique Using Population-based (Sero)Surveillance
Brief Title: Characterising Transmission of SARS-CoV-2 in a Peri-urban Population in Mozambique
Acronym: AfriCoVER
Status: Completed | Type: Observational
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); Instituto Nacional de Saúde, Mozambique (Other Government); Institut de Recherche pour le Developpement (Other Government); UMC Utrecht (Other)
Responsible Party: Sponsor
Other Study IDs: AfriCoVER
Record Dates: First submitted 2020-06-16; First posted 2020-06-22 (Actual); Results first posted 2025-01-22 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Nasal swabs (for all possible Covid-19cases)
  * Dried Blood Spots (only in a subset of the population, 2400 individuals)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A population-based COVID19 surveillance in a household cohort will be set-up using an existing Household demographic surveillance system (HDSS). From any individual in this population with any respiratory symptom or loss of smell or taste, with or without fever, investigators will collect a respiratory specimen and test these for SARS-CoV-2 virus, during 12 months. Demographic, epidemiological and clinical data of possible cases and of the source population will be recorded at baseline.

An age-stratified serial sero-survey will be conducted at baseline in a subset of the population in the population-based COVID19 surveillance, and at 3, 6 and 12 months, after confirmation of community transmission.

DETAILED DESCRIPTION:
The investigators will use the established HDSS to set up population-based COVID19 surveillance in a household cohort. From any individual in this population with any respiratory symptom or loss of smell or taste, with or without fever, investigators will collect a respiratory specimen and test these for SARS-CoV-2 virus by PCR, during 12 months. These cases will be identified through bi-weekly household visits, through an alert system involving community leaders and HDSS interviewers, or when presenting with symptoms at healthcare centres or the referral hospital. Demographic, epidemiological and clinical data (comorbidities, medication, obesity, HIV, TB, smoking) of possible cases and of the source population will be recorded at baseline; recent illness, potential risk exposure of each household member (including duration and type) to SARS-CoV-2 positive individuals, uptake of measures to reduce exposure/transmission, and barriers to the uptake of such measures, will be recorded/updated during every household visit.

An age-stratified serial sero-survey will be conducted at baseline in a subset of the population in the population-based COVID19 surveillance, and at 3, 6 and 12 months, after confirmation of community transmission.

ELIGIBILITY:
Inclusion Criteria:

* Any individual enrolled in the Polana Caniço-HDSS: All members residing in the household for at least 3 months (infants, children, adults, elderly), regardless of age, underlying conditions, medical history, infection or disease status or history
* Able and willing to provide written informed consent: by the household head for the surveillance; by each selected participant for the sero-survey.

No Exclusion Criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The Polana Caniço-HDSS (Health- and Demographic Surveillance System) has been established since 2017. In total, 2108 households (defined as residents of the same building, sharing a cooking area) have been enrolled in the HDSS. All members residing in the household for at least 3 months (infants, children, adults, elderly) are enrolled in the HDSS.
  All households in the HDSS (2108 during the last round, in 2019) consenting to participate in the study will be visited biweekly by a trained HDSS interviewer, following the same procedures as in routine HDSS rounds, specified in the HDSS protocol (Instituto Nacional de Saude, 2016). We assume the same number of households will consent to participate as in other HDSS rounds.
Sampling Method: Non-Probability Sample
Enrollment: 6049 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2022-03-29 (Actual); Study Completion 2022-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc-Alain Widdowson, Dr, Principal Investigator — Institute of Tropical Medicine
Locations (1):
- INS, Maputo, Mozambique

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During December 2020-March 2022, households of a population cohort in Polana Caniço, Maputo, Mozambique, were visited or phoned biweekly. Residents reporting any respiratory sign, anosmia, or ageusia, was asked to self-administer a nasal swab, for SARS-CoV-2 PCR testing. Of a subset of 1400 participants, dried blood spots were repeatedly collected, three-monthly, from fingerpicks at home.
Groups:
- All Participants Visited: During 11925 household visits in 1561 households 6049 participants were covered
Period: Overall Study
Arm/Group | All Participants Visited
Started | 6049
Participants Undergoing a Nasal Swab | 579
Participants Undergoing Dry Blood Spot Collection | 1412
Completed | 6049
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort Participants: Screened/visited Participants, not having self-reported first confirmed COVID-19 episodes
Arm/Group | Cohort Participants
Number analyzed (Participants) | 6049
Age, Customized [Count of Participants; unit: Participants]
  0-9 years | 1331
  10-19 years | 1570
  20-29 years | 1128
  30-39 years | 644
  40-49 years | 519
  50-59 years | 406
  60-69 years | 318
  ≥70 years | 133
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3245
  Male | 2804
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Socio-economic quintile [Count of Participants; unit: Participants]
  Lowest | 836
  Low | 1015
  Med | 1063
  Med/high | 1078
  highest | 1132
  unknown | 925
Education [Count of Participants; unit: Participants]
  none | 88
  primary | 2646
  secondary | 1735
  higher | 277
  unknown | 1303
Health worker Reported comorbidities [Count of Participants; unit: Participants]
  reported comorbidities | 196
  no reported comorbidities | 5853
BMI [Count of Participants; unit: Participants]
  underweight | 817
  normal | 802
  overweight | 281
  obesity | 237
  unknown | 3912
Smoking [Count of Participants; unit: Participants]
  Non smoker | 5738
  (ex) smoker | 251
  unknown | 60
Public transportation [Count of Participants; unit: Participants]
  None | 3948
  bus/train | 2013
  moto taxi/shared taxi | 19
  unknown | 69
Sharing bedroom [Count of Participants; unit: Participants]
  1-2 pers. | 3311
  3 or more pers. | 2646
  unknown | 92
Sharing toilet with other household [Count of Participants; unit: Participants]
  sharing toilet | 896
  no sharing toilet or not recorded | 5153
Handwash facility [Count of Participants; unit: Participants]
  sink/faucet | 1748
  bucket/jar/kettle | 1204
  none | 3005
  unknown | 92
Water available in house [Count of Participants; unit: Participants]
  Yes | 2153
  no | 3804
  unknown | 92

OUTCOME MEASURES:

1. Primary Outcome: COVID-19 Disease Incidence Rate (Symptomatic Infections Per Month)
Description: Estimate the COVID-19 incidence rate over a 12 month period in peri-urban Maputo
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: infections per 1000 person-years
Groups:
- Persons Followed up: During 11925 household visits in 1561 households, covering 6049 participants
Arm/Group | Persons Followed up
Number analyzed (Participants) | 6049
infections per 1000 person-years | 364.5 [352.8 to 376.1]

2. Primary Outcome: COVID-19 Related Hospitalization Rate Due to SARS-CoV-2
Description: Estimate the hospitalization rate related to SARS-CoV-2 over a 12 month period in peri-urban Maputo
Time Frame: 12 months
Population: confirmed COVID-19 cases followed up at day 28
Measure: Count of Participants; unit: Participants
Groups:
- Confirmed COVID-19 Cases: confirmed COVID-19 cases
Arm/Group | Confirmed COVID-19 Cases
Number analyzed (Participants) | 85
Participants | 0

3. Primary Outcome: Case (Disease) Fatality Risk (Percent) Due to SARS-CoV-2
Description: Estimate the COVID-19 case fatality of cases detected during a 12 month period in peri-urban Maputo.
  A part of the cases (92) was followed up until 28 days, a part (54) until 56 days.
Time Frame: 12 months
Population: 92 confirmed cases followed up after 28 days, of whom 54 again after 56 days
Measure: Count of Participants; unit: Participants
Arm/Group | Confirmed COVID-19 Cases
Number analyzed (Participants) | 92
Participants | 1

4. Primary Outcome: Percentage Asymptomatic Infections
Description: Estimate the percentage of infections that are asymptomatic.This percentage is not available by age group. The percentage comes from combining 2 measures: the incidence rates (per age groups) with the overal incidence rate of SARS-CoV-2 infection in the first 6 months of the study, inferred from the change in sero-prevalence
Time Frame: 12 months
Measure: Number; unit: percentage of infections
Arm/Group | Confirmed COVID-19 Cases
Number analyzed (Participants) | 85
percentage of infections | 86.6

5. Primary Outcome: Percentagge of Participants With SARS-CoV-2 Infection Annually
Description: Estimate the attack rate of SARS-CoV-2 infection during 6 months in peri-urban Maputo. Crude sero-prevalence among study participants.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Participants Dry Blood Spot: Of a subset of 1400 participants, dried blood spots were repeatedly collected, three-monthly, from fingerpicks at home.
Arm/Group | Participants Dry Blood Spot
Number analyzed (Participants) | 1412
percentage of participants
  in December 2020 | 4.8 [1.1 to 8.6]
  in June 2021, when 3.0% of participants was vaccinated with at least one dose of vaccine | 34.7 [20.2 to 49.3]

ADVERSE EVENTS:
Time Frame: As there is no investigational product in this study, adverse events were not monitored/assessed. Death was followed up in COVID cases for 56 days.
Description: As there is no investigational product in this study, adverse events were not monitored/assessed.
Groups:
- All Participants Visited: all participants that were visited throughout the study
Arm/Group | All Participants Visited
All-Cause Mortality (participants affected / at risk) | 1/92
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-14): https://cdn.clinicaltrials.gov/large-docs/65/NCT04442165/Prot_SAP_000.pdf